CLINICAL TRIAL: NCT03573154
Title: Nicotine Pharmacokinetic Study and Volatile Organic Compound Analysis in Exhaled Breath After Electronic Cigarette Utilization.
Brief Title: Nicotine Pharmacokinetic in Blood and Analysis of Exhaled Breath After E-cigarette Smoking.
Acronym: VAPexp'Air
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 6911
Record Dates: First submitted 2018-04-11; First posted 2018-06-29 (Actual); Last update posted 2021-12-23 (Actual); Status verified 2021-12

CONDITIONS: Electronic Cigarette
Keywords: nicotine; e-cigarette; exhaled breath; pharmacokinetic model
MeSH Terms: conditions — Vaping

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- e-liquid 1 (Other)
  Interventions: Other: administration of the liquid 1 and then the liquid 2
- e-liquid 2 (Other)
  Interventions: Other: administration of the liquid 2 and then the liquid 1

INTERVENTIONS:
Other: administration of the liquid 1 and then the liquid 2 — The patient will received the e-liquid 1 in the first visit and the e-liquid 2 in the second
  Arms: e-liquid 1
Other: administration of the liquid 2 and then the liquid 1 — The patient will received the e-liquid 2 in the first visit and the e-liquid 1 in the second
  Arms: e-liquid 2

SUMMARY:
Electronic or e-cigarettes are battery-powered devices that deliver vapor which may be inhaled in the manner tobacco is smoked. The e-liquid is usually a solution containing propylene glycol and/or vegetable glycerin, nicotine, and flavor concentrates, although some e-liquids also are sold as non-nicotine containing products. The long- and short-term public health consequences of e-cigarette use, including the effects of e-cigarettes on tobacco use behavior, are not well understood. However, the prevalence of e-cigarette use appears to be undergoing a rapid increase.

In this study the investigators propose to analyze nicotine pharmacokinetic in blood and to compare the exhaled breath before and after e-cigarette smoking. They want to obtain a pharmacokinetic model of this population for nicotine. And they want to identify if molecules contained in vapor are absorbed, metabolized or modified by the organism.

ELIGIBILITY:
Inclusion Criteria:

* Subject who has already used electronic cigarette
* Subject who has been using electronic cigarette for more than one month and/or Tobacco smoker (traditional cigarettes)
* Subject without history of chronic pathology
* Subject not taking long-term drug treatment
* Subject able to understand studie's aims and risk

Exclusion Criteria:

* Subject with a chronic respiratory pathology
* Subject suffering from a respiratory or acute otorhinolaryngology pathology in progress or recent
* Subject under alcohol withdrawal
* Subject with heavy drinking or daily use of illegal drugs
* Subject with epilepsy
* Subject having hypersensitivity to one of the compounds of the spraying liquid
* Subject with liver failure
* Subject with severe renal impairment (GFR <60 ml / min)
* Subject with an allergy to the molecules contained in the e-liquid
* Subject suffering from claustrophobia
* Pregnancy or breastfeeding

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-12-19 (Actual); Primary Completion 2022-06-15 (Estimated); Study Completion 2022-08-03 (Estimated)

PRIMARY OUTCOMES:
Concentration of nicotine in blood at Baseline | At T0 (during the nicotine's absorption by the patient)
  Concentration of nicotine in blood made by liquid chromatography/mass spectrometry method.
Concentration of nicotine in blood at 10 minutes | At T10 min after the nicotine's absorption
  Concentration of nicotine in blood made by liquid chromatography/mass spectrometry method.
Concentration of nicotine in blood at 20 min | At T20 min after the nicotine's absorption
  Concentration of nicotine in blood made by liquid chromatography/mass spectrometry method.
Concentration of nicotine in blood at 40 min | At T40 min after the nicotine's absorption
  Concentration of nicotine in blood made by liquid chromatography/mass spectrometry method.
Concentration of nicotine in blood at 80 min | At T80 min after the nicotine's absorption
  Concentration of nicotine in blood made by liquid chromatography/mass spectrometry method.

CONTACTS AND LOCATIONS:
Locations (1):
- Hopitaux Universitaires de Strasbours, Strasbourg, Grand Est, France